CLINICAL TRIAL: NCT01839747
Title: Evaluation of PET/MRI in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael Gee, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-307
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hematologic Malignancy
Keywords: Pediatric
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging (Experimental): PET-MRI PET-CT
  Interventions: Procedure: PET-MRI; Procedure: PET-CT

INTERVENTIONS:
Procedure: PET-MRI — Imaging
Procedure: PET-CT — Imaging

SUMMARY:
This research study is a Pilot study (a small preliminary study to assess the feasibility of a larger, more in depth study involving a new test or procedure) and is being done to evaluate the feasibility and accuracy of PET/MRI in the evaluation of cancer. PET/MRI is a FDA approved technology that is currently being studied to assess its accuracy and utility in the diagnosis and management of a variety of diseases and patient populations. The focus of this particular study will be to compare the performance of PET/MRI in its ability to detect and characterize cancerous tumors using positron emission topography and computed tomography (PET/CT) as a reference standard.

DETAILED DESCRIPTION:
If you agree to participate in this study you will be asked to fill out a screening questionnaire to determine if you can participate. No additional screening tests or procedures will be necessary prior to your participation in this study.

If the screening questionnaire shows that you are eligible to participate in the research study, you will be scheduled to undergo your PET/MRI in conjunction with your PET/CT. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

After th screening procedures confirm that you are eligible to participate in the research study:

1. You will schedule your PET/CT examination with the MGH radiology department according to the orders and instructions of your oncologist (cancer doctor)
2. Study personnel will coordinate the scheduling of your PET/MRI examination to coincide with date and time of your PET/CT examination
3. Following the performance of your PET/CT examination you will be transported (with your accompanying family member(s)) to the Charlestown Navy Yard MGH imaging facility where you will undergo your PET/MRI examination. No additional dose of radioactive tracer (a substance which is labeled with a radioactive molecule that can be tracked within your body based on the radiation it emits) will be given as part of your PET/MRI examination
4. The PET/MRI will take up to 60 minutes to complete and after it is completed you will be free to go
5. The PET/MRI images will be interpreted by physicians (trained radiologists) as part of the study analysis; however no report of the findings will be made available to you. You will have access to the results of the PET/CT examination as you would any other clinical imaging examination.
6. If you are willing, with each subsequent PET/CT examination you undergo while enrolled in the study, you will also undergo a PET/MRI examination
7. The study will last for 12 months, after which time you will no longer be enrolled

ELIGIBILITY:
Inclusion Criteria:

* Able to lie comfortably on a bed inside the scanner for 60 minutes as assessed by physical examination and medical history

Exclusion Criteria:

* Requirement for sedation or anesthesia of any kind in order to undergo MRI scanning
* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing
* Pregnancy or breastfeeding
* Pre-existing medical conditions or claustrophobic reactions, and any greater than normal potential for cardiac arrest

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of Imaging Quality between PET-MRI and PET-CT | 2 years
  To perform a qualitative comparison of image quality between PET-MRI and PET-CT exams being performed on pediatric oncology patients during the same visit

SECONDARY OUTCOMES:
Comparison of PET-MRI SUV Values and PET-CT FDG Reference | 2 years
  To compare the ability of PET-MRI to determine the extent of active malignancy by comparing PET-MRI SUV values with PET-CT FDG reference
Assessment of Unexpected Indeterminate Lesions | 2 years
  To assess the number of unexpected indeterminate lesions detected on PET-MRI and PET-CT studies requiring additional workup

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gee, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States